CLINICAL TRIAL: NCT03817931
Title: Higher Neural and Cognitive Changes Following Anticholinergic Versus Beta 3 Agonist Versus Placebo Treatments in Female Patients With Overactive Bladder: a Multicenter Randomized Controlled Pilot Trial
Brief Title: Higher Neural Changes Following Anticholinergic, Beta 3 Agonist, or Placebo in Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: The Methodist Hospital Research Institute (Other); International Urogynecological Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 160362
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2019-08

CONDITIONS: Overactive Bladder; Dementia; Lower Urinary Tract Symptoms; Incontinence, Urge
MeSH Terms: conditions — Urinary Bladder, Overactive; Dementia; Lower Urinary Tract Symptoms; Urinary Incontinence, Urge | interventions — Cholinergic Antagonists; Solifenacin Succinate; Adrenergic beta-3 Receptor Agonists; mirabegron; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Permuted block stratified by recruitment site
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization using a random number system will be performed by the compounding pharmacy. Records linking subject number to their allocation will be kept by the pharmacy, inaccessible to the investigator, patient, care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo pill identical will be identical to tablets in the other 2 arms.
  Interventions: Diagnostic Test: Functional magnetic resonance imaging (fMRI); Diagnostic Test: Rey Auditory Verbal Learning Test (RAVLT)
- Anticholinergic (Active Comparator): Solifenacin 5 mg tablet orally once daily for 30 days
  Interventions: Drug: Anticholinergic; Diagnostic Test: Functional magnetic resonance imaging (fMRI); Diagnostic Test: Rey Auditory Verbal Learning Test (RAVLT)
- Beta-3 agonists, adrenergic (Active Comparator): Mirabegron 25 mg tablet orally once daily for 30 days
  Interventions: Drug: Beta-3 Agonists, Adrenergic; Diagnostic Test: Functional magnetic resonance imaging (fMRI); Diagnostic Test: Rey Auditory Verbal Learning Test (RAVLT)

INTERVENTIONS:
Drug: Anticholinergic — Tablet taken once daily.
  Other Names: Solifenacin; VESIcare
  Arms: Anticholinergic
Drug: Beta-3 Agonists, Adrenergic — Tablet taken once daily.
  Other Names: Mirabegron; Myrbetriq
  Arms: Beta-3 agonists, adrenergic
Diagnostic Test: Functional magnetic resonance imaging (fMRI) — All subjects have fMRI at baseline and again after 30 days
Diagnostic Test: Rey Auditory Verbal Learning Test (RAVLT) — All subjects have RAVLT at baseline and again after 30 days. RAVLT evaluates: short-term auditory-verbal memory, rate of learning, learning strategies, retroactive, and proactive interference, presence of confabulation of confusion in memory processes, retention of information, and differences between learning and retrieval.
  Other Names: cognitive testing

SUMMARY:
Women presenting with overactive bladder symptoms will be randomized to one of 3 arms (anticholinergic, beta-3 agonist, placebo). They will undergo baseline cognitive testing, functional MRI of the brain. Cognitive testing and functional MRI will be repeated after taking their double blinded intervention for 30 days.

DETAILED DESCRIPTION:
Women presenting to the urology clinic with complaints of urinary urgency, frequency in the absence of urinary tract infection or other obvious pathology will be screened for inclusion/exclusion criteria. Qualifying subjects will be consented.

Baseline health information, bladder symptom questionnaires (Overactive Bladder-questionnaire(OABq), Patient Perception of Bladder Condition (PPBC)), Personal Health Questionnaire-9 (PHQ-9),Hamilton Anxiety Rating Scale (HAM-A), Montreal cognitive assessment (MoCA) will be given. If baseline depression (PHQ-9 score 15 or greater),dementia (MoCA score 25 or less), anxiety (HAM-A score 25-30) are noted the subject is excluded. 15 patients will be recruited from Baylor Scott & White Health Urology clinic, and 15 patients will be recruited from Houston Methodist Urology clinic.

They will schedule a date within 1 month for the Rey Auditory Verbal Learning Test (RAVLT) and brain functional MRI (fMRI). RAVLT test is performed, followed by resting state fMRI and memory task during fMRI. Vials of medication will be distributed. Vials will be labeled 1-30 and will contain 30 tablets each. The anticholinergic and beta-3 agonist tablets will be encapsulated to look identical to the placebo tablet. Subjects will be reimbursed at this visit. fMRI images at baseline and post-intervention will be analyzed by a radiologist for incidental findings.

One week and two weeks after initiating their tablets, phone interviews will inquire about pill count, side effects, and any new medications. Follow up testing date will be scheduled during the call. The same questions will be repeated at completion of the tablets (30 days after initiation).

At completion of the tablets, subjects return to Houston Methodist for repeat RAVLT and fMRI. Subjects will be reimbursed the other half of their compensation at this visit.

An expert physicist will analyze the BOLD signal intensity and FC pattern in a priori selected regions of interest before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of age 50 to 90 years old with OAB as defined by the International Continence Society (Urgency with or without urge incontinence, usually with frequency and nocturia in the absence of urinary tract infection or other obvious pathology) who report that symptoms cause moderate problems using the PPBC.
* English-speaking and able to consent

Exclusion Criteria:

* Males are excluded to eliminate prostate pathology and urethral strictures, as well as possible bias of gender differences on fMRI.
* Subjects with moderately severe or severe depression (screening score of 15 or more) on the Personal Health Questionnaire-9 (PHQ-9)
* Subjects with moderate to severe anxiety (screening score 25-30) on the Hamilton Anxiety Rating Scale (HAM-A)
* A screening score indicating below normal cognitive function at baseline (score of 25 or less) on the montreal cognitive assessment.
* Subjects with neurologic disorders, dementia, prior cerebrovascular accident, neurogenic bladder or post-void residual greater than 250 mL
* Anticholinergics for OAB or beta 3 agonists use for treatment of OAB in the preceding six months prior to enrollment
* Pregnant or planning to become pregnant in the next six months, or current breastfeeding
* The inability to undergo MRI

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Functional connectivity on MRI | 29 +/-1 days
  Functional connectivity during a word recognition task will be compared within subjects from baseline and after 29+/- 1 day of intervention medication.
Resting state blood oxygenation level dependent (BOLD)changes | 29 +/-1 days
  During resting state, BOLD changes will be compared within subjects from baseline and after 29+/- 1 day of intervention medication.
Diffusion tensor imaging | 29 +/-1 days
  Fractional anisotropy and mean diffusivity from diffusion tensor images will be compared within subjects from baseline and after 29+/- 1 day of intervention medication.

SECONDARY OUTCOMES:
Score on Rey Auditory Verbal Learning Test (RAVLT) | 30 days
  Baseline testing will be compared with post-intervention testing
Overactive bladder questionnaire (OAB-q) | 30 days
  Baseline score of this validated questionnaire will be compared with post-intervention score
Patient Perception of Bladder Condition (PPBC) | 30 days
  Baseline score of this validated questionnaire will be compared with post-intervention score

CONTACTS AND LOCATIONS:
Overall Officials: Jill Danford, MD, Principal Investigator — Baylor Scott and White Health; Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute; Rachel High, DO, Principal Investigator — Baylor Scott and White Health
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott and White Health, Temple, Texas

IPD SHARING:
Plan to Share IPD: No
There is not a plan.

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Houston Methodist Translational Imaging Center — https://www.houstonmethodist.org/research/our-research/cores/translational-imaging-core-facilities/